CLINICAL TRIAL: NCT05032352
Title: Predictive Assay for Decision Making in Adjuvant Therapy (PADMA)
Brief Title: Predictive Assay for Decision Making in Adjuvant Therapy
Acronym: PADMA
Status: Terminated | Type: Observational
Why Stopped: Non-safety related, reallocation of resources
Sponsor: Insight Molecular Diagnostics (Industry)
Collaborators: ClinLogix. LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: PADMA Trial
Record Dates: First submitted 2021-08-26; First posted 2021-09-02 (Actual); Last update posted 2022-11-14 (Actual); Status verified 2021-09

CONDITIONS: Carcinoma, Non-Small-Cell Lung
Keywords: Non-squamous Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Adjuvants, Pharmaceutic; Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Treatment Arm: Treatment Arm 1: 4 cycles of adjuvant treatment with a standard NSCLC cisplatin-based doublet regimen or carboplatin-based regimen of physician choice.
  Treatment 1A: other adjuvant therapy or combination of adjuvant therapies (targeted therapy, immunotherapy, or other)
  Interventions: Drug: Adjuvant; Other: Observation
- Observation only: All patients will be observed for progression free survival and overall survival to the end of study or death, whichever occurs first.
  Interventions: Other: Observation

INTERVENTIONS:
Drug: Adjuvant — Adjuvant treatment with a standard NSCLC platin-based doublet, 4 cycle (21-day) regimen of the investigator's choice (Arm 1) or other adjuvant therapy (Arm 1a) which can include combination of chemotherapy and targeted therapy, immunotherapy or other.
  Groups: Treatment Arm
Other: Observation — All patients will be observed for progression free survival and overall survival to the end of study or death, whichever occurs first.

SUMMARY:
Prospective Registrational Trial to Define Real World Outcomes of Patients with Completely Resected Stage I or IIA (tumor < or = 5cm, node negative) Non-squamous Non-Small Lung Cancer (NSCLC) Identified as High, Intermediate, or Low Risk by a 14-Gene Prognostic Assay DetermaRx being Considered for Adjuvant Platinum-based chemotherapy or other adjuvant therapy versus Observation

DETAILED DESCRIPTION:
This is a prospective, non-randomized, 2 arm, multi-center study in patients with histologically documented non-squamous NSCLC who have undergone complete resection (R0) of the primary tumor with pathologically stage I or IIA disease. Routine paraffin-embedded tumor specimens from completely resected (R0) stage I or IIA patients with non-squamous NSCLC will undergo testing with the DetermaRx 14-Gene Prognostic Assay and will be designated as HIGH, INTERMEDIATE or LOW risk by the assay. The physician and patient will determine the best treatment course and will be assigned to treatment arm based on decision of adjuvant therapy or observation:

1. Adjuvant treatment with a standard NSCLC platin-based doublet, 4 cycle (21-day) regimen of the investigator's choice (Arm 1) or other adjuvant therapy (Arm 1a) which can include combination of chemotherapy and targeted therapy, immunotherapy or other.
2. Observation (Arm 2) All patients will be observed for progression free survival and overall survival to the end of study or death, whichever occurs first.

All patients will be observed for disease free survival and overall survival to the end of study or death, whichever occurs first

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent using the appropriate approved Institutional Review Board (IRB) approved consent.
2. Age ≥ 18 years
3. Able to comply with the protocol, including acceptable candidacy for adjuvant chemotherapy and likely compliance with follow-up for anticipated length of study (18 months from randomization).
4. Adequate tissue sample, paraffin block with tumor occupying at least 25% of the tissue surface area, for the 14 -gene prognostic assay, DetermaRx
5. Histologically documented completely resected (R0) Stage I or IIA non-squamous NSCLC per 8th edition, TNM staging system. Mixed histology cases (adenosquamous), large cell, or adenocarcinoma not otherwise classified (NOS) are eligible for the study, as long as they contain at least some component that is neither squamous cell, nor small cell nor neuroendocrine. Eligible resections include lobectomy, bilobectomy, segmentectomy, sleeve lobectomy and pneumonectomy. Resections via segmentectomy or wedge resection should be limited to patients with a peripheral tumor 2 cm or less with wide margins (> 2 cm or > the size of the nodule). Complete resection must also be accompanied, at a minimum, by intra-operative systematic mediastinal lymph node sampling. Systematic sampling is defined as removal of at least one representative lymph node each from levels 4 and 7 for a right-sided cancer and from levels 5 and/or 6 and 7 for left-sided cancers. Complete mediastinal lymph node dissection (MLND), however, is preferred, and is defined as resection of all lymph nodes at those same levels for right- and left-sided cancers.
6. ECOG performance status 0-1
7. No prior anti-neoplastic (NSCLC ) treatment in the pre-operative or post-operative setting (including chemotherapy, targeted therapy, immunotherapy, radiation, ablative procedures, etc.)

Exclusion Criteria:

1. Final pathologic diagnosis of pure squamous cell, pure small cell, or pure neuroendocrine histology, or any combination of only these three histological subtypes.
2. Evidence of greater than stage IIA pathologic staging
3. Evidence of incomplete resection (R1)
4. Prior systemic chemotherapy or anti-cancer agent for NSCLC
5. Any pre- or post-operative radiotherapy for the index tumor being considered for enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with non-squamous NSCLC who have undergone complete resection (R0) of the primary tumor and who have been documented to have pathologically confirmed stage I or IIA disease
Sampling Method: Probability Sample
Enrollment: 55 (Actual)
Dates: Start 2022-01-28 (Actual); Primary Completion 2022-10-28 (Actual); Study Completion 2022-10-28 (Actual)

PRIMARY OUTCOMES:
Free Survival (DFS) | 30-36 months
  To compare Disease Free Survival (DFS) in patients with resected, stage I or IIA non-squamous NSCLC found to be at HIGH/INTERMEDIATE Risk by DetermaRX choosing to undergo adjuvant therapy using a platinum-based doublet or other adjuvant therapy versus observation.

SECONDARY OUTCOMES:
Secondary Objectives | 30-36 months
  1. To evaluate use patterns of DetermaRx in guiding use of adjuvant platinum-based chemotherapy across early-stage resected lung cancer
  2. To evaluate DFS in DetermaRx LOW risk patients who are put on observation alone
  3. To evaluate whether use of DetermaRx HIGH/INTERMEDIATE vs. LOW to guide adjuvant platinum-based therapy results in improved OS in patients
  4. To evaluate if EGFR mutational status impacts use of adjuvant platinum-based therapy in DetermaRx HIGH/INTERMEDIATE vs. LOW patients

OTHER OUTCOMES:
Exploratory Analyses | 30-36 months
  1. To evaluate predictive value of DetermaRx in driver positive NSCLC patients receiving chemotherapy, targeted therapy or both.
  2. To evaluate predictive value of DetermaRx early NSCLC patients receiving chemotherapy + immunotherapy or other combination adjuvant therapies
  3. To evaluate predictive value of other histological features on pathology in association with DetermaRx as well as additional biomarkers (i.e., KRAS, TP53, STK11, PD-L1 expression, etc.) if performed by physician in combination with DetermaRx results and related outcomes

CONTACTS AND LOCATIONS:
Overall Officials: Corey Langer, MD, Principal Investigator
Locations (18):
- United States (18):
  - City of Hope National Medical Center, Duarte, California
  - MedStar Washington Hospital Center, Washington D.C., District of Columbia
  - George Washington Medical Faculty Associates, Washington D.C., District of Columbia
  - Jupiter Medical Center, Jupiter, Florida
  - Piedmont Cancer Center, Atlanta, Georgia
  - Northshore University Healthsystem, Evanston, Illinois
  - The University of Kansas Hospital, Kansas City, Kansas
  - Our Lady of the Lake Regional Medical Center, Baton Rouge, Louisiana
  - Penn Presbyterian Medical Center, Philadelphia, Pennsylvania
  - Texas Oncology-San Antonio Medical Center, San Antonio, Texas
  - Methodist Healthcare, San Antonio, Texas
  - Texas Oncology-Wichita Falls Cancer Center, Wichita Falls, Texas
  - Virginia Cancer Specialists, Fairfax, Virginia
  - Mary Washington Hospital, Fredericksburg, Virginia
  - Providence Regional Medical Center Everett, Everett, Washington
  - Peace Health, Vancouver, Washington
  - West Virginia University Medicine, Morgantown, West Virginia
  - Medical College of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: Undecided
Not determined yet

REFERENCES:
- [Result] Wu YL, Tsuboi M, He J, John T, Grohe C, Majem M, Goldman JW, Laktionov K, Kim SW, Kato T, Vu HV, Lu S, Lee KY, Akewanlop C, Yu CJ, de Marinis F, Bonanno L, Domine M, Shepherd FA, Zeng L, Hodge R, Atasoy A, Rukazenkov Y, Herbst RS; ADAURA Investigators. Osimertinib in Resected EGFR-Mutated Non-Small-Cell Lung Cancer. N Engl J Med. 2020 Oct 29;383(18):1711-1723. doi: 10.1056/NEJMoa2027071. Epub 2020 Sep 19. PMID 32955177